CLINICAL TRIAL: NCT01910246
Title: Cardiovascular Effects of Metformin on Obesity With Subclinical Myocardial Dysfunction
Brief Title: Cardiovascular Effects of Metformin on Obesity
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No funding
Sponsor: University of California, San Francisco (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MetforminMRI; Cardiac MRI Metformin; Metformin Cardiac MRI (Other: UCSF)
Record Dates: First submitted 2013-04-22; First posted 2013-07-29 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Insulin Resistance
Keywords: Metformin; Insulin Resistance; Cardiac Function
MeSH Terms: conditions — Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin, Insulin Resistance, Cardiac Function, (Experimental): Metformin Hydrochloride Tablets will be administered with a start dose of 500mg twice daily with meals.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
It has been shown that asymptomatic obese adolescents can demonstrate abnormal regional myocardial contraction, with preserved global cardiac function. Metformin has been shown to decrease cardiovascular mortality in patients with type 2 diabetes and insulin resistance, but the mechanism of cardiovascular protection is unknown.

The purpose of this study is to evaluate the reversibility of subclinical cardiovascular abnormalities in obese adolescents with insulin resistance after a six-month course of Metformin. The investigators hypothesized that the beneficial effects of Metformin will be progressive and sustained after six months of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents 12 to 17 years old under clinical care at the UCSF WATCH clinic
* Body mass index> 95th percentile for age and gender according to the Centers for Disease Control and Prevention 2000 growth charts for the United States
* Insulin resistant after 6 months of healthy diet and exercise
* Able to understand the assent form

Exclusion Criteria:

* Patients with known cardiac disease
* Patients with contraindications to metformin as listed below:

  * Renal disease or renal (serum creatinine levels ≥1.5 mg/dL for males, and ≥1.4 mg/dL for females;
  * Known hypersensitivity to Metformin;
  * Acute or chronic metabolic acidosis;
* Patients with contraindications to MRI including:

  * Cardiac pacemaker;
  * Claustrophobia;
  * Metallic foreign body in the eye,
  * Aneurysm clip in the brain
* Pregnancy;
* Patients who could not stay still for 30 minutes within the MRI scanner due to other reasons besides claustrophobia

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Circumferential Strain change after a six-month course of Metformin. | 6 months
  Circumferential strain will be measured by cardiac MRI before and after the treatment. Change in circumferential strain (measured as percentage from end-diastolic wall thickness) from baseline is the main outcome of this study. We hypothesize that abnormal baseline circumferential stain will increase and reach normal values after Metformin treatment. We hypothesized that the beneficial effects of Metformin will be progressive and sustained.

CONTACTS AND LOCATIONS:
Overall Officials: Karen G Ordovas, MD, MAS, Principal Investigator — University of California, San Francisco; David Saloner, PhD, Study Director — University of California, San Francisco
Locations (1):
- UCSF, Radiology and Biomedical Imaging, San Francisco, California, United States